CLINICAL TRIAL: NCT04233385
Title: Pain and Immobility After Breast Cancer Surgery: A Community-Based Randomized Controlled Trial of Myofascial Massage Treatment
Brief Title: Myofascial Massage for Pain and Immobility Following Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Ash Sehgal, Co-Director Center for Reducing Health Disparities, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB18-00912
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Mastectomy; Lymphedema; Pain, Shoulder; Mobility Limitation
Keywords: breast cancer; breast surgery; myofascial massage; shoulder immobility
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Shoulder Pain; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: A blinded research assistant will perform all outcomes assessments of objective functional measures. Participants will be told they are being randomized into two different types of massage, however, we will not refer to they myofascial massage as "intervention" or the light touch as "active control"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myofascial Massage (Experimental): Participants randomized to this group will receive 30 minutes of myofascial massage to their affected breast, chest, and shoulder areas twice a week for 2 months. Therapists will follow a detailed 8 week protocol developed with a massage therapy consultant and the study team.
  Interventions: Other: Myofascial Massage
- Light Touch (Active Comparator): Participants randomized to this group will receive 30 minutes of light touch to their affected breast, chest, and shoulder areas twice a week for 2 months.
  Interventions: Other: Light Touch

INTERVENTIONS:
Other: Myofascial Massage — The myofascial protocol outlines techniques, areas of the body, as well as time to be spent for each technique for a total of 25 minutes. The remaining 5 minutes of the massage are for the massage therapist to tailor myofascial massage to the needs and circumstances of each participant. In order to provide some level of customization, the therapist will determine the impact of massage on the participant's pre-existing pain and/or mobility limitations. Second, the therapist will assess the soft tissues around the affected breast, chest, and shoulder to determine the locations of pain, tissue firmness, and restricted mobility. Third, the therapist will use effleurage and petrissage techniques to gently massage the identified locations to soften and release the tissues. Techniques used will include deep friction of muscles, sustained compression, and fascial stretch.
  Arms: Myofascial Massage
Other: Light Touch — Participants randomized to this group will receive 30 minutes of light touch to their affected breast, chest, and shoulder areas twice a week for 2 months. Therapists will follow a detailed light touch protocol for each of the 16 sessions. In addition, the therapist will inquire about the participant's response to the previous light touch treatment. Second, the therapist will assess the soft tissues around the affected breast, chest, and shoulder to determine the locations of pain, tissue firmness, and restricted mobility. Third, the therapist will place both hands on the participant for 3 minutes at each identified location. Pressure will be very light and consistent, with no side-to-side movement.
  Arms: Light Touch

SUMMARY:
About 25-50% of women who undergo breast cancer surgery develop persistent chest wall pain and shoulder mobility limitations following surgery. The pain and mobility limitations adversely affect quality of life, sleep, and body image. Unfortunately, current treatments for pain and mobility limitations have variable efficacy. Based on a review of relevant pre-, intra-, and post-operative factors, investigators reasoned that myofascial massage may address contributors to pain and mobility limitations following breast cancer surgery. Investigators propose a randomized controlled trial looking at myofascial massage compared to a light touch group to look at the effects on pain and immobility following breast cancer surgery.

DETAILED DESCRIPTION:
Myofascial massage is a deep tissue massage that focuses on muscles as well as the connective tissue that surrounds muscles, bones, and ligaments. The study team subsequently conducted a pilot randomized controlled trial involving 21 women with persistent pain and mobility limitations many months after surgery. They found that women who received myofascial massage to the affected breast/chest/shoulder had marked reductions in pain and mobility limitations and significant improvements in quality of life compared to a control group who received relaxation massage. They also established a practice-based research network of over 50 northeast Ohio massage therapists to guide future work.

The study team now proposes a full scale randomized controlled trial involving 202 women with persistent pain and mobility limitations at 2 participating sites. To help differentiate between the specific effects of myofascial massage and non-specific effects due to prolonged touch and attention from a massage therapist, the study will include an active control group that will receive light touch. Participants in each group will receive 30 minutes of treatment twice weekly for 2 months. Primary analyses will determine the impact of myofascial massage on pain and mobility limitations. Secondary analyses will examine the impact of myofascial massage on a number of secondary outcomes, including range of motion, quality of life, sleep, and body image.

Innovative features of the proposed project include a rigorous randomized controlled trial design, inclusion of an active control group, direct targeting of the affected breast/chest/shoulder, assessment of multiple mechanistic and patient-centered outcomes, and involvement of a massage practice-based research network. Investigators anticipate that the project will lead to a new and effective approach for addressing a major source of morbidity for women with breast cancer. Furthermore, the project may serve as a model for future trials of manual therapy among individuals with chronic medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Female
* Undergone breast cancer surgery 3-18 months ago
* Completed all treatment for breast cancer within the last 18 months (i.e. radiation, IV chemotherapy, surgery)
* Not expected to have any additional surgery (i.e. planning for reconstruction)
* Self reported chronic pain or immobility since surgery

Exclusion Criteria:

* Under age 18
* Not female
* Surgery < 3 months ago
* End all cancer treatments (surgery, radiation, chemotherapy) > 18 months ago
* Presence of lymphedema
* Open wounds or sores
* Currently on anticoagulants
* Currently receiving massage treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is limited to females who have undergone breast cancer surgery.
Enrollment: 132 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in self reported pain scores | Baseline, 1 month, 2 months, 8 months, and 14 months
  Shoulder Pain and Disability Index "SPADI", 5 pain items rated on a 10 point likert scale, where 0 is no pain at all and 10 is the worst pain imaginable
Change in self reported mobility scores | Baseline, 1 month, 2 months, 8 months, and 14 months
  Shoulder Pain and Disability Index "SPADI", 8 mobility items rated on a 10 point likert scale, where 0 means no issues with mobility and 10 means they are unable to complete the task

SECONDARY OUTCOMES:
Range of Motion | Baseline, 2 months, 14 months
  Shoulder range of motion measured by goniometer and objective functional tasks
Pressure/Pain Threshold | Baseline, 2 months, 14 months
  Pressure to pain threshold as measured by algometer
Grip Strength | Baseline, 2 months, 14 months
  Hand grip strength measured by dynamometer
Tissue Flexibility | Baseline, 2 months, 14 months
  Change in tissue flexibility as measured by adherometer
Quality of Life Survey-Functional Assessment of Cancer Therapy - Breast (FACT-B) | Baseline, 2 months, 14 months
  44-item questionnaire designed to measure physical well-being, social/family well-being, emotional well-being, functional well-being, and additional breast cancer-specific concerns

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Ewertz M, Jensen AB. Late effects of breast cancer treatment and potentials for rehabilitation. Acta Oncol. 2011 Feb;50(2):187-93. doi: 10.3109/0284186X.2010.533190. PMID 21231780
- [Background] Hayes SC, Johansson K, Stout NL, Prosnitz R, Armer JM, Gabram S, Schmitz KH. Upper-body morbidity after breast cancer: incidence and evidence for evaluation, prevention, and management within a prospective surveillance model of care. Cancer. 2012 Apr 15;118(8 Suppl):2237-49. doi: 10.1002/cncr.27467. PMID 22488698
- [Background] Hidding JT, Beurskens CH, van der Wees PJ, van Laarhoven HW, Nijhuis-van der Sanden MW. Treatment related impairments in arm and shoulder in patients with breast cancer: a systematic review. PLoS One. 2014 May 9;9(5):e96748. doi: 10.1371/journal.pone.0096748. eCollection 2014. PMID 24816774
- [Background] Thomas-Maclean RL, Hack T, Kwan W, Towers A, Miedema B, Tilley A. Arm morbidity and disability after breast cancer: new directions for care. Oncol Nurs Forum. 2008 Jan;35(1):65-71. doi: 10.1188/08.ONF.65-71. PMID 18192154
- [Background] Johansen S, Fossa K, Nesvold IL, Malinen E, Fossa SD. Arm and shoulder morbidity following surgery and radiotherapy for breast cancer. Acta Oncol. 2014 Apr;53(4):521-9. doi: 10.3109/0284186X.2014.880512. Epub 2014 Feb 5. PMID 24495044
- [Background] Meretoja TJ, Leidenius MHK, Tasmuth T, Sipila R, Kalso E. Pain at 12 months after surgery for breast cancer. JAMA. 2014 Jan 1;311(1):90-92. doi: 10.1001/jama.2013.278795. No abstract available. PMID 24381969
- [Background] Colagiuri B, Christensen S, Jensen AB, Price MA, Butow PN, Zachariae R. Prevalence and predictors of sleep difficulty in a national cohort of women with primary breast cancer three to four months postsurgery. J Pain Symptom Manage. 2011 Nov;42(5):710-20. doi: 10.1016/j.jpainsymman.2011.02.012. Epub 2011 May 26. PMID 21620648
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841